CLINICAL TRIAL: NCT01281228
Title: The Effect of GLP-1 Receptor Activation on Central Reward and Satiety Circuits in Response to Food Stimuli in Obesity and Diabetes
Brief Title: The Effect of GLP-1 Receptor Activation on Central Reward and Satiety in Obesity and Diabetes
Acronym: Braini-Ex
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: Eli Lilly and Company (Industry); Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, RG IJzerman, Dr., Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: DC2010Exbrain001; 2010-023635-42 (EudraCT Number)
Record Dates: First submitted 2011-01-20; First posted 2011-01-21 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2015-06

CONDITIONS: Diabetes Mellitus; Diabetes Mellitus, Type 2; Obesity
Keywords: Exenatide; Type 2 diabetes mellitus; Incretin hormones; GLP-1 agonist; Satiety; Reward
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2; Obesity | interventions — Exenatide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- exenatide (Experimental): Infusion of exenatide; loading dose 50 ng/min during 30 min, followed by a maintenance dose 20ng/min for the rest of the tests.
  Interventions: Drug: exenatide
- exenatide + exendin (9-39) (Experimental): exenatide infusion: loading dose 50 ng/min during 30 min, followed by a maintenance dose 20 ng/min for the rest of the test. And infusion of exendin(9-39) 600pM/kg/min.
  Interventions: Drug: exenatide + exendin (9-39)
- saline (Placebo Comparator): saline infusion, with the same infusion speed
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: exenatide — The loading dose is 50 ng/min during 30 min, followed by a maintenance dose 20 ng/min for the rest of the tests.
  Other Names: Byetta
  Arms: exenatide
Drug: exenatide + exendin (9-39) — The loading dose is 50 ng/min during 30 min, followed by a maintenance dose 20 ng/min for the rest of the tests. Exendin 9-39 will be infused intravenously at doses of 600 pM/kg • min.
  Arms: exenatide + exendin (9-39)
Drug: placebo — saline infusion
  Arms: saline

SUMMARY:
Glucagon-like peptide 1 (GLP-1) based therapies, such as exenatide, are already successfully employed in the treatment of Type 2 Diabetes (T2DM). Exenatide improves glycemic control and is associated with reduced food intake and body weight. The investigators hypothesize that it affects central reward and satiety circuits and that this may contribute to the weight loss.

DETAILED DESCRIPTION:
The aim of the project is to determine 1) whether GLP-1 receptor activation of CNS reward and satiety circuits occurs, in the context of food(-related) stimuli; if this effect is altered in obese and diabetic compared to lean individuals 2) if it is independent of other postprandial metabolic and hormonal changes 3) if this effect is GLP-1-receptor-mediated 4) if the CNS changes correlate with subsequent feeding behaviour.

Methods The investigators will compare 16 obese T2DM-patients, 16 normoglycemic obese and 16 healthy lean individuals, with respect to food(-related) neuronal activity in central reward and satiety circuits by blood oxygen level-dependent (BOLD) fMRI. fMRI will be performed during intravenous infusion of a) the GLP-1 receptor agonist exenatide; b) exenatide and a GLP-1 receptor antagonist (exendin 9-39)(to investigate whether the exenatide-induced effects are GLP-1-receptor mediated) or c) saline; in randomized order, on separate days. To tease out concomitant postprandial metabolic and hormonal influences, measurements will be performed during a somatostatin pancreatic clamp with replacement of basal insulin, glucagon and growth hormone. Finally, to correlate changes in brain activity with subsequent feeding behavior, the investigators will measure food intake, self-reported hunger, satiety and mood, during a choice-buffet after the scanning.

Expected Results This project will gain insight into (CNS) mechanisms underlying the observed effects of the GLP-1 receptor agonist exenatide on food intake and body weight in obese, diabetic and healthy lean individuals. These findings may increase our understanding of the development of obesity and weight loss problems in obese and diabetic individuals and the role of GLP-1 in the central regulation of feeding behavior/appetite control.

ELIGIBILITY:
Inclusion Criteria:

For all 3 study groups:

1. age 18-70 years.
2. Men and women. For women, only postmenopausal women (as ascertained by serum FSH) will be included in order to avoid variations related to the menstrual cycle.
3. To promote comparability and to overcome the interference of lateralization, only right-handed persons will be included.

For the healthy lean subjects, inclusion criteria will be:

1. body-mass index (BMI) of <25 kg/m2
2. stable bodyweight (<5% reported change during the previous 3 months)
3. Normal fasting and 2-h postload glucose as ascertained during a 75-g oral glucose tolerance test (OGTT)

For the normoglycemic obese individuals, inclusion criteria will be:

1. body-mass index (BMI) ≥30 kg/m2
2. stable bodyweight (<5% reported change during the previous 3 months)
3. Normal fasting and 2-h postload glucose as ascertained during a 75-g oral glucose tolerance test (OGTT)

For the obese T2DM individuals, inclusion criteria will be:

1. Diagnosed with T2DM (20) > 3 months prior to screening
2. BMI ≥30 kg/m2
3. HbA1c 6.2-8.5%
4. Treatment with metformin at a stable dose for at least 3 months.

Exclusion Criteria:

In the obese T2DM patients, no blood glucose- and weight lowering agents will be allowed within 3 months before screening except for metformin. The normoglycemic lean and obese individuals will not be allowed to take blood glucose-lowering agents at any time before and during the study.

For all individuals, exclusion criteria will be:

1. congestive heart failure (NYHA II-IV)
2. chronic renal failure (glomerular filtration rate < 60 mL/min/1.73m2 per Modification of Diet in Renal Disease (MDRD)) or serious liver impairment
3. a history of gastrointestinal disorders, including gastroparesis, pancreatitis and cholelithiasis
4. neurological illness
5. malignancy
6. pregnancy or breast feeding
7. implantable devices
8. substance abuse
9. addiction
10. contra-indication for MRI, such as claustrophobia or pacemaker
11. any psychiatric illness, including eating disorders and depression
12. hypersensitivity to the active substance or to any of the excipients
13. chronic use of glucocorticoids or centrally acting drugs within 2 weeks immediately prior to screening
14. use of cytostatic or immuno-modulatory agents
15. participation in other studies
16. individuals who have received treatment within the last 30 days with a drug that has not received regulatory approval for any indication at the time of study entry
17. individuals who are investigator site personnel directly affiliated with the study, or are immediate family of investigator site personnel directly affiliated with the study. Immediate family is defined as a spouse, parent, child, or sibling, whether biological or legally adopted
18. individuals who have previously completed or withdrawn from this study or any other study investigating GLP-1 receptor agonist or dipeptidyl peptidase (DPP)-4 within 6 months
19. individuals, who in the opinion of the investigator, are unsuitable in any other way to participate in this study
20. individuals who are employed by Amylin Pharmaceutical Inc. or Eli Lilly & company (that is, employees, temporary contract workers, or designees responsible for conducting the study). Immediate family of Amylin or Lilly employees may participate in sponsored clinical trials, but are not permitted to participate at an Amylin or Lilly facility. Immediate family is defined as a spouse, parent, child, or sibling, whether biological or legally adopted
21. poor commandment of the Dutch language or any (mental) disorder that precludes full understanding the purpose, instruction and hence participation in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2011-09; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Differences in neuronal activity in CNS reward and satiety circuits | 1 hour
  Differences in neuronal activity in CNS reward and satiety circuits (including striatum, amygdala, orbitofrontal cortex, insula, hypothalamus), as represented by BOLD fMRI signal change from baseline (%) in response to food(-related) stimuli, between obese T2DM patients, normoglycemic obese individuals and normoglycemic healthy lean subjects.

SECONDARY OUTCOMES:
Feeding behavior | 2 hours
  Feeding behavior, measured as quantitative (kcal) and qualitative (energy density as well as nutrient composition; carbohydrate/fat/protein) changes in food choice during a choice-buffet lunch, will be compared between groups and conditions.
Self-reported hunger | 2 hours
  Self-reported hunger, satiety, fullness and prospective food consumption, will be rated on 100 mm visual analogue scales before and after the meal.

CONTACTS AND LOCATIONS:
Overall Officials: Michaela Diamant, MD PhD, Principal Investigator — VU University Medical Center, Diabetes Center
Locations (1):
- VU University Medical Center, Amsterdam, De Boelelaan 1117, Netherlands

REFERENCES:
- [Derived] van Bloemendaal L, IJzerman RG, Ten Kulve JS, Barkhof F, Konrad RJ, Drent ML, Veltman DJ, Diamant M. GLP-1 receptor activation modulates appetite- and reward-related brain areas in humans. Diabetes. 2014 Dec;63(12):4186-96. doi: 10.2337/db14-0849. Epub 2014 Jul 28. PMID 25071023